# **Evaluation of Preventive (Stay Safe) Training Program of Child Abuse for Teachers and Children: A Randomized Controlled Trial from Multan City**

**Informed consent** 

By

Zainab Noor Hussain
PSY-07
M.Phil. Applied Psychology

**Supervisor** 

Dr. Rizwana Amin



**Department of Applied Psychology** 

Bahauddin Zakariya University, Multan

**Informed Consent Form for children** 

Date: September 15, 2018

Name of Principal Investigator: Zainab Noor Hussain

This Informed Consent Form has two parts:

• Information Sheet (to share information about the research with you)

• Certificate of Consent (for signatures if you agree to take part)

You will be given a copy of the full Informed Consent Form

**PART I: Information Sheet** 

Introduction

I am zainab, working on the prevention of child abuse. Child abuse is common in Pakistan now a day, every child have a risk of being abused. This research study work on the prevention of children from abuse, if you find this information healthy then allow your child to participate in this study.

**Purpose** 

The purpose of this research is to give children knowledge about abuse and safe them from this dangerous issue. This research provide information to children related to the prevention of child abuse and give them learning about the safety skills.

**Type of Research Intervention** 

The research intervention consist of training as children receive training of safety skills by the use of programme named "stay safe programme"

**Participant selection** 

Children of class 1 and 2 are the participants of the study. Children are selected form schools where whole class of 1 and 2 is included.

**Voluntary Participation** 

Child participation in this research is entirely voluntary. It is your choice whether to participate or not. If child is not feel comfortable in the study he or she will withdrawal from research at any time.

**Procedures and Protocol** 

The procedure of the study is as follows:

**B.** Description of the Process

Stay safe programme is used in this research where children receive training about the safety skills which include good touch and bad touch, bullying, secrets, bribes, safe and unsafe events,

etc. this is lesson based from which covers 5 to 6 topics related to the safety skills of children about abuse.

#### Duration

The duration of the programme would be 2 weeks and then after 1 week participants again participate to describe how much they understand the lessons by answer the questions in the scales.

### **Side Effects**

It does not have any side effects as it is beneficial completely.

#### **Benefits**

If child participate in the study they are able to defend themselves even when are all alone. It is beneficial for them.

## **Confidentiality**

It is informed you that all the information of participants kept confidential and use in research purpose only. Participants name, age, etc. would be secure and used safely only in study.

## Right to Refuse or Withdraw

It is participant duty if he or she is feasible to continue the study and receive complete training. If participant feel uncomfortable, he or she allows to leave or withdrawal from research at any time.

#### Who to Contact

If participant have any questions participant may ask them now or later, even after the study has started. If you wish to ask questions later, you may contact any of the following: [Zainab Noor Hussain,

+923078686352,

zainabnoorhussain@gmail.com]

**PART II: Certificate of Consent** 

I have been invited to participate in research of child abuse. I understand that it will involve

beneficial and have lessons related to prevention of abuse. I am aware that there may be some

benefit to me personally. I have been provided with the name of a researcher who can be

easily contacted using the number and address I was given for that person.

I have read the foregoing information, or it has been read to me. I have had the opportunity to

ask questions about it and any questions that I have asked have been answered to my

satisfaction. I consent voluntarily to participate as a participant in this research and understand

that I have the right to withdraw from the research at any time.

Signature of child's parent:

(Participant name is kept confidential)

Name of Researcher: Zainab Noor Hussain